CLINICAL TRIAL: NCT03144648
Title: Molecular Subtypes of Premenopausal Breast Cancer in Latin American Women (PRECAMA): a Multicenter Population-based Case-control Study
Brief Title: PRECAMA: Molecular Subtypes of Premenopausal Breast Cancer in Latin American Women
Acronym: PRECAMA
Status: Recruiting | Type: Observational
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: University of Chile (Other); Fundación Inciensa (Other); Instituto Nacional de Salud Publica, Mexico (Other); Universidad de Antioquia (Other); Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PRECAMA
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum, plasma, red blood cells, buffy coats, urine, and for cases, DNA from tumor tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Incident primary invasive breast cancer cases aged 20-45 years are recruited from major cancer hospitals in five Latin American cities (Barretos, Mexico City, San Jose, Medellin, and Santiago) prior to any treatments. For each subject, complete questionnaire data on socio-demographic factors, health and reproductive history, early risk factors, physical activity, diet, environmental risk factors, ethnicity, and family history of cancer are collected. Validated and standardized food frequency questionnaires are administered to gather information on diet. Anthropometry is measured according to standardized protocols. Blood and urine samples are also collected for biomarker analyses. Highly standardized immunohistochemical and molecular analyses are performed to identify cancer subtypes
  Interventions: Other: lifestyle
- Controls: Women with no cancer recruited from the population residing in the same cities for at least 3 years and matched to cases on age (+/- 5 years) and health care institution. For each subject, complete questionnaire data on socio-demographic factors, health and reproductive history, early risk factors, physical activity, diet, occupation, environmental risk factors, ethnicity, and family history of cancer are collected. Validated and standardized food frequency questionnaires are administered to gather information on diet. Anthropometry is measured according to standardized protocols. Blood and urine samples are also collected for biomarker analyses.
  Interventions: Other: lifestyle

INTERVENTIONS:
Other: lifestyle — Observational study

SUMMARY:
Breast cancer has become a major public health problem in Latin America, as it is the most common form of cancer among women. Women are more likely to develop breast cancer at younger age, and to be diagnosed at an advanced stage compared to western women. Over the past twenty years, the mortality from breast cancer in Latin America has also been increasing very rapidly, and is currently the leading cause of cancer mortality. Little is known on specific risk factors for premenopausal breast cancer in general, and in Latin America in particular. There is a lack of specific knowledge on tumor molecular and pathological characteristics of breast cancer in Latin America premenopausal women, and this has major consequences on cancer treatment and survival.

To improve our understanding on determinants of breast cancer incidence and mortality in young Latin America women and support preventive actions, we implemented an international, population-based multi-center study in Latin America: the PRECAMA study (Molecular Subtypes of Premenopausal Breast Cancer in Latin American Women (PRECAMA): a multicenter population-based case-control study).

PRECAMA is coordinated by the International Agency for Research on Cancer (IARC), and is conducted within 4 Latin American countries: Mexico, Costa Rica, Colombia and Chile. Major aims of the project are the following:

1. To develop a multi-centric population-based case-control study on breast cancer in premenopausal women in several countries in Latin America with structured collection of individual, clinical, pathological information and biological specimens, according to strictly controlled protocols
2. To characterize, in these populations, the subtypes of premenopausal breast cancer on the basis of their molecular and pathological phenotypes
3. To improve the identification of specific endogenous/exogenous factors, and disentangle the interplay of these different factors with regard to breast tumor subtypes.
4. Provide advanced training, induce a structuring effect on the breast cancer research community in Latin America and influence the public health agenda regarding the management of breast cancer.

The results of our study will be of utmost importance to understand the etiology of breast cancer in Latin America countries, and would provide important information on the role of modifiable exposures for breast cancer prevention.

DETAILED DESCRIPTION:
Breast cancer (BC) has become a major public health problem in Latin America (LA), as it is the most common form of cancer among women. In Women are more likely to develop BC at younger age, and to be diagnosed at an advanced stage compared to western women. Over the past twenty years, the mortality from BC in LA has also been increasing very rapidly, and is currently the leading cause of cancer mortality among LA women. The large number of incident BC cases among premenopausal women, which is only partly explained by the population age-structure, is therefore of major concern. Little is known on specific risk factors for premenopausal BC in general, and in LA in particular, and risk factors related to diet, obesity and low physical activity play a role on incidence and mortality. Estrogen receptor (ER) and/or Progesterone receptor (PR) expression in breast tumors may differ according to risk factors and to molecular pathological characteristics. There is a lack of specific knowledge on tumor molecular and pathological characteristics of BC in premenopausal women, particularly in lower resource countries where the hormone-dependence status is poorly documented. This has major consequences on cancer treatment and survival.

To improve our understanding of determinants of BC incidence and mortality in young Latin America women and support preventive actions, we implemented an international, population-based multi-center case-control study in LA: the PRECAMA study (Molecular Subtypes of Premenopausal Breast Cancer in Latin American Women (PRECAMA): a multicenter population-based case-control study).

PRECAMA is coordinated by the International Agency for Research on Cancer (IARC), and is conducted within 4 Latin American countries: Mexico, Costa Rica, Colombia and Chile. Major aims of the project are the following:

1. To develop a multi-centric population-based case-control study on BC in premenopausal women in several countries in LA with structured collection of individual, clinical, pathological information and biological specimens, according to strictly controlled protocols
2. To characterize, in these populations, the subtypes of premenopausal BC on the basis of their molecular and pathological phenotypes
3. To improve the identification of specific endogenous/exogenous factors, and disentangle the interplay of these different factors with regard to breast tumor subtypes.
4. Provide advanced training, induce a structuring effect on the BC research community in LA and influence the public health agenda regarding the management of BC.

Standardized methods and questionnaires have been developed and implemented as well as standard operating procedures for laboratory activities. Incident primary invasive cases aged 20-45 years are recruited from major cancer hospitals in four large Latin American cities (Mexico City, San Jose, Medellin, and Santiago) prior to any treatments. Controls for the study are selected from the population residing in the same cities for at least 3 years and matched to cases on age (+/- 5 years) and health care institution. For each subject, complete questionnaire data on socio-demographic factors, health history, reproductive history, use of hormones, early risk factors, body silhouette at different ages, physical activity, diet, occupation, environmental risk factors, ethnicity, and family history of cancer are collected. Validated and standardized food frequency questionnaires are administered to gather information on diet. Anthropometry (body weight, standing and sitting height, waist and hip circumferences) are measured according to standardized protocols. Blood and urine samples are also collected for biomarker analyses. For all cases, highly standardized immunohistochemical and molecular analyses are performed to identify BC subtypes.

The results of our study will be of utmost importance to understand the etiology of breast cancer in Latin America countries in epidemiological transition, and would provide important information on the role of modifiable exposures on the disease which may provide important support for breast cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* woman between 20 and 45 years old
* woman less than 3 years older or younger than the case
* living in the area that the study is taking place during the past 3 years
* woman menstruated at least once in the past 12 months
* woman diagnosed with a primary breast cancer by histopathological examination (only for cases)

Exclusion Criteria:

* woman receiving tumor treatment, such as radiotherapy, chemotherapy or anti-estrogens (for example, tamoxifen) (except treatment for non-melanoma skin cancers)
* woman taking (or has previously taken) any of the following medications in the past 6 months: tamoxifen, Evista (raloxifene), Fareston (toremifene), Aromasin (exemestane), Femara (letrozole), Arimidez (anastrozole) or Megace (megestrol)
* woman suffering from chronic kidney failure
* woman having a pathology that will hinder adequate communication
* woman who is pregnant or nursing
* woman who has been previously diagnosed with a cancer(except for non-melanoma skin cancers)
* any other reason to exclude

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal Latin America women
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-10-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
breast cancer | at recruitment
  breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Rinaldi, PhD, Principal Investigator — International Agency for Research on Cancer, Lyon, France; Maria Luisa Garmendia, PhD, Principal Investigator — INTA, Universidad de Chile, Santiago, Chile; Carolina Porras, PhD, Principal Investigator — Proyecto Epidemiológico Guanacaste, Fundación INCIENSA, Costa Rica; Gabriela Torres-Mejía, PhD, Principal Investigator — Instituto Nacional de Salud Pública, Cuernavaca, Mexico; Gloria I Sánchez, PhD, Principal Investigator — Grupo Infección y Cáncer, Universidad de Antioquía, Medellín, Colombia; Fabiana Vazquez, Principal Investigator — Barretos Cancer Hospital
Locations (13):
- Barretos Cancer Hospital, Barretos, Brazil
- Chile (3):
  - INC, Santiago, Independencia
  - Hso-Crsco, Santiago, Peñalolén
  - FALP, Santiago, Providencia
- Colombia (7):
  - Grupo Infección y Cáncer. Universidad de Antioquia, Medellín, Antioquia
  - International Hospital of Colombia, Bucaramanga, Bucaramanga
  - Facultad de Medicina, Universidad del Norte, Barranquilla
  - Hospital Internacional de Colombia Fundacion Cardiovascular de Colombia, Bucaramanga
  - SENOSAMA foundation, Bucaramanga
  - Instituto de Oncología HematoOncologos, Cali
  - Public Health University of Narino, Pasto
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), San José, Provincia de San José, Costa Rica
- Instituto Nacional de Salud Pública (INSP), Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://precama.iarc.fr